CLINICAL TRIAL: NCT01018173
Title: A Randomized Double Blind, Placebo-controlled Clinical Trial to Assess the Effects of Taspoglutide (RO5073031) on Cardiovascular Outcomes in Subjects With Inadequately Controlled Type 2 Diabetes and Established Cardiovascular Disease
Brief Title: A Study of Taspoglutide in Patients With Inadequately Controlled Diabetes Mellitus Type 2 and Cardiovascular Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NC25113; 2009-014986-22
Record Dates: First submitted 2009-11-20; First posted 2009-11-23 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — taspoglutide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Drug: placebo
- taspoglutide (Experimental)
  Interventions: Drug: taspoglutide

INTERVENTIONS:
Drug: placebo — sc weekly
  Arms: placebo
Drug: taspoglutide — 10 mg sc weekly for 4 weeks, followed by 20 mg sc weekly
  Arms: taspoglutide

SUMMARY:
This randomized, double-blind, placebo-controlled parallel arm study will assess efficacy and safety and the effects of taspoglutide on cardiovascular events in patients with inadequately controlled type 2 diabetes mellitus and established cardiovascular disease. Patients will be randomized to receive either taspoglutide subcutaneously (sc) 10mg weekly for 4 weeks followed by 20mg sc weekly, or weekly sc placebo, in addition to background anti-hyperglycemic medication and standard of care treatment for cardiovascular disease. Anticipated time on study treatment is up to 2 years. Target sample size is 2000 patients.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >18 years of age
* diabetes mellitus type 2
* HbA1c >/=6.5% and </=10% at screening
* BMI >/=23kg/m2
* cardiovascular disease with onset >/=1 month prior to screening

Exclusion Criteria:

* diagnosis or history of type 1 diabetes or secondary forms of diabetes
* acute metabolic diabetic complications within past 6 months
* severe hypoglycemia </=1 month prior to screening
* clinically significant gastrointestinal disease
* history of chronic or acute pancreatitis
* current New York Heart Association (NYHA) class IV heart failure or post-transplantation cardiomyopathy
* severely impaired renal function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2118 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Time to cardiovascular composite primary endpoints | event-driven, cardiovascular assessments weeks 1,4,12 and every 3 to 4 months thereafter

SECONDARY OUTCOMES:
Secondary cardiovascular composite endpoints | event-driven, cardiovascular assessments weeks 1,4,12 and every 3 to 4 months thereafter
Individual components of primary cardiovascular composite endpoints | event-driven, cardiovascular assessments weeks 1,4,12 and every 3 to 4 months thereafter
Total mortality | assessed at end of study, week 104
Metabolic and renal function parameters: HbA1c, fasting plasma glucose, body weight, lipid profile, albumin/creatinine ratio (ACR), albuminuria, glomerular filtration rate (GFR) | laboratory assessments weeks 4 and 12, and every 3 to 6 months thereafter

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (234):
- United States (70):
  - Phoenix, Arizona
  - Tucson, Arizona
  - Buena Park, California
  - Calabasas, California
  - Fresno, California
  - Santa Ana, California
  - Walnut Creek, California
  - Centennial, Colorado
  - Colorado Springs, Colorado
  - Trumbull, Connecticut
  - Washington D.C., District of Columbia
  - Clearwater, Florida
  - Delray Beach, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Ponte Verde, Florida
  - Bloomingdale, Illinois
  - Chicago, Illinois
  - Evansville, Indiana
  - Baltimore, Maryland
  - Oxon Hill, Maryland
  - Jackson, Mississippi
  - St Louis, Missouri
  - North Platte, Nebraska
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Nashua, New Hampshire
  - Toms River, New Jersey
  - Mineola, New York
  - New York, New York
  - Calabash, North Carolina
  - Cary, North Carolina
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Mooresville, North Carolina
  - Raleigh, North Carolina
  - Bismarck, North Dakota
  - Cleveland, Ohio
  - Kettering, Ohio
  - Toledo, Ohio
  - Bend, Oregon
  - Medford, Oregon
  - Portland, Oregon
  - Beaver, Pennsylvania
  - Levittown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pottstown, Pennsylvania
  - Greer, South Carolina
  - Hickory Grove, South Carolina
  - Bristol, Tennessee
  - Johnson City, Tennessee
  - Austin, Texas
  - Carrollton, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Irving, Texas
  - North Richland Hills, Texas
  - Richardson, Texas
  - San Antonio, Texas
  - Temple, Texas
  - Salt Lake City, Utah
  - Burke, Virginia
  - Hampton, Virginia
  - Manassas, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Winchester, Virginia
  - Tacoma, Washington
- Australia (4):
  - Freemantle, Queensland
  - Herston, Queensland
  - Elizabeth Vale, South Australia
  - Melbourne, Victoria
- Brazil (4):
  - Fortaleza, Ceará
  - Campina Grande do Sul, Paraná
  - Rio de Janeiro, Rio de Janeiro
  - São Paulo, São Paulo
- Bulgaria (5):
  - Byala
  - Pleven
  - Plovdiv
  - Sofia
  - Varna
- Canada (4):
  - Barrie, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Sherbrooke, Quebec
- Czechia (12):
  - Havířov
  - Jindřichův Hradec
  - Mariánské Lázně
  - Olomouc
  - Pardubice
  - Prague
  - Rakovník
  - Ricany U Prahy
  - Semily
  - Trutnov
  - Uherské Hradiště
  - Ústí nad Labem
- Denmark (4):
  - Aalborg
  - Ballerup Municipality
  - Hvidovre
  - Vejle
- Estonia (6):
  - Paide
  - Saku
  - Tallinn
  - Tartu
  - Viljandimaa
  - Võru
- Germany (11):
  - Bad Lauterberg im Harz
  - Bad Oeynhausen
  - Bochum
  - Dortmund
  - Dresden
  - Essen
  - Hamburg
  - Kleve
  - Neuss
  - Nuremberg
  - Wuppertal
- Hungary (11):
  - Balatonfüred
  - Budapest
  - Debrecen
  - Gyula
  - Hódmezővásárhely
  - Komárom
  - Makó
  - Sopron
  - Szikszó
  - Úrhida
  - Veszprém
- India (15):
  - Ahmedabad
  - Aurangabad
  - Bangalore
  - Banglore
  - Bhopal
  - Chennai
  - Hyderabad
  - Jaipur
  - Kochi
  - Kolkata
  - Madurai
  - Mangalore
  - Mumbai
  - Nagpur
  - Pune
- Jerusalem, Israel
- Lithuania (5):
  - Alytus
  - Kaunas
  - Klaipėda
  - Panevezys
  - Vilnius
- Malaysia (3):
  - George Town
  - Johor Bahru
  - Kelantan
- Mexico (10):
  - Aguascalientes
  - Chihuahua City
  - Cuernavaca
  - Culiacán
  - Durango
  - Juarez, Distrito Federal
  - Mexico City
  - México
  - Monterrey
  - Tampico
- Poland (12):
  - Gdansk
  - Gdynia
  - Kamieniec Ząbkowicki
  - Katowice
  - Kielce
  - Krakow
  - Lodz
  - Poznan
  - Płock
  - Radom
  - Warsaw
  - Wroclaw
- Romania (9):
  - Bacau
  - Baia Mare
  - Bucharest
  - Constanța
  - Galati
  - Oradea
  - Ploieşti
  - Târgu Mureş
  - Timișoara
- Russia (6):
  - Barnaul
  - Kemerovo
  - Moscow
  - Novosibirsk
  - S. Petersburg
  - Saint Petersburg
- Slovakia (8):
  - Banská Bystrica
  - Bratislava
  - Dolný Kubín
  - Komárno
  - Levice
  - Lučenec
  - Prievidza
  - Trenčín
- South Africa (8):
  - Cape Town
  - Durban
  - Johannesburg
  - Observatory, Cape Town
  - Port Elizabeth
  - Pretoria
  - Richards Bay
  - Soweto
- Spain (2):
  - Lugo, Lugo
  - Madrid, Madrid
- Taiwan (3):
  - Taichung
  - Taipei
  - Taoyuan
- Thailand (2):
  - Bangkok
  - Chiang Mai
- Ukraine (8):
  - Kharkiv
  - Kiev
  - Lviv
  - Mykolaiv
  - Poltava
  - Ternopil
  - Vinnitsa
  - Zaporizhzhya
- United Kingdom (11):
  - Bexhill-on-Sea
  - Birmingham
  - Cardiff
  - Chorley
  - Dundee
  - Glasgow
  - Liverpool
  - London
  - Manchester
  - Reading
  - Salford